CLINICAL TRIAL: NCT03446768
Title: Monitoring and Peer Support to Improve Treatment Adherence and Outcomes in Patients With Overlap Chronic Obstructive Pulmonary Disease and Sleep Apnea Via a Large PCORnet Collaboration
Brief Title: Monitoring and Peer Support to Improve Treatment Adherence and Outcomes
Acronym: O2VERLAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: COPD Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20173014
Record Dates: First submitted 2018-01-15; First posted 2018-02-27 (Actual); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Obstructive Sleep Apnea
Keywords: COPD; OSA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reactive Care (RC) (Active Comparator): Participants in the RC arm of the study will be provided access to the COPD Information Line if they feel they would benefit from the support of a peer health coach. Peer health coaches working the information line are patients also living with COPD who can offer peer level support.
  Interventions: Other: Peer support
- Proactive Care (PC) (Active Comparator): Participants in the PC arm of the study will be provided access to the COPD Information Line if they feel they would benefit from the support of a peer health coach. Peer health coaches working the information line are patients also living with COPD who can offer peer level support. Additionally, the PC group will also receive access to an online study portal which houses an educational health curriculum covering topics related to COPD and OSA. The portal allows participants to send online messages to peer coaches and respiratory therapist coaches. PC group will also receive weekly updates.
  Interventions: Other: Peer support; Other: Online platform; Other: Respiratory Therapist support

INTERVENTIONS:
Other: Peer support — Access to educational and informational support by a trained peer coach
Other: Online platform — An online platform that provides educational, informational and access to several therapeutic device metrics
  Arms: Proactive Care (PC)
Other: Respiratory Therapist support — Limited medical support provided by trained Respiratory Therapists.
  Arms: Proactive Care (PC)

SUMMARY:
The O2VERLAP study investigators would like to find out if individuals living with both COPD and OSA would benefit from an online, educational curriculum, coupled with access to peer support (i.e. telephone and online chatting with peers) and remote CPAP adherence monitoring data. The curriculum and peer coaching is meant to provide participants the information and tools they need to be more compliant in using their CPAP device.

DETAILED DESCRIPTION:
The O2VERLAP study focuses on a subset of the Chronic Obstructive Pulmonary Disease (i.e. COPD) community that are also living with a diagnosis of Sleep Apnea (i.e. SA); having a diagnosis of both COPD and SA is referred to as Overlap Syndrome (i.e. OS). There are about 300 million people living with COPD globally; of those, OSA affects 17% of adults and over 25% of older adults with rates increasing in association with the obesity epidemic. So, there are approximately 51-75 million individuals living with OS worldwide. This subset of the COPD community is met with increased morbidity and mortality rates compared to either diagnosis alone. The primary treatment for OSA is continuous positive airway pressure (i.e. CPAP, sometimes shortened to PAP).

When individuals with OS are adherent to their nighttime CPAP therapies they see significantly improved outcomes, comparable to individuals living with a diagnosis of COPD alone. As a result, the primary aim of this study is to improve CPAP adherence in patients living with OS. The study investigators hope to do this through a proactive, peer-support based intervention, supplemented by an online curriculum and access to remote CPAP adherence monitoring data. Peer-coaches will include individuals who are living with COPD and OSA, who are similar to the study population. The COPD Information Line associates will act in this peer- support role through dyadic, telephone-based communication and through secure online chat. The COPD Information Line peer-coaches will be able to provide participants experience- based advice, patient-centered guidance on troubleshooting adherence barriers, as well as patient-centered advice on how to facilitate CPAP adherence. Peer coaches will also include Respiratory Therapists who will be able to provide coaching from the perspective of a caregiver. Additionally, all peer based support aims to provide emotional and social support to participants. The participants will have the ability to chat with their peer coaches online, both in real-time and asynchronously, and will additionally have weekly check ins with their coaches. The curriculum addresses many common CPAP adherence barriers and facilitators. The investigators hope that the combination of peer-support and self-learning will cultivate patient activation, self-management strategies and improve participant's health literacy. Ultimately, the investigators expect that this will improve CPAP adherence rates at 6 weeks and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: >40 years
* Primary language: English
* Diagnosed with both Chronic Obstructive Pulmonary Disease (COPD) and Obstructive Sleep Apnea (OSA)
* Prescription for positive airway pressure therapy (PAP). There should be no minimum or maximum flow required (i.e., no limitation on PAP modality).
* Access to the internet viand a PC, tablet, or smart phone to complete all study activities from home or remotely
* PAP device with wireless modem

Exclusion Criteria:

* Non-English speakers
* Life expectancy less than or equal to six months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Stepnowsky, PhD, Principal Investigator — University of California, San Diego; Elisha Malanga, BS, Principal Investigator — COPD Foundation
Locations (1):
- COPD Foundation Inc., Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reactive Care (RC) | Proactive Care (PC)
Started | 141 | 153
Completed | 141 | 152
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reactive Care (RC) | Proactive Care (PC) | Total
Number analyzed (Participants) | 141 | 153 | 294
Age, Continuous [Mean (Full Range); unit: years] | 64.7 [45 to 86] | 64.2 [41 to 89] | 64.4 [41 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 68 | 139
  Male | 70 | 85 | 155
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 128 | 132 | 260
  Race: Black or African American | 6 | 10 | 16
  Race: Multiple Race | 6 | 7 | 13
  Race: Asian | 1 | 0 | 1
  Race: Other | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 141 | 153 | 294

OUTCOME MEASURES:

1. Primary Outcome: Change in CPAP Adherence at 6 Weeks
Description: CPAP adherence is being measured through remote adherence monitoring of all participants; the study inclusion criteria requires all participants be using a CPAP device with wireless modem, the wireless modem allows the study investigators to accurately measure participants CPAP usage daily. Participants CPAP device record the 'total time connected' each day or total time the device is being used (i.e. units are hours per day). Study investigators will retroactively access and collect 30-days of baseline adherence data, prior to randomization, to measure the participants level of baseline adherence. The study investigators will then track participants total time using their CPAP device in hours, each day, for the duration of the participants enrollment (i.e. about three months).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: hours per night of CPAP use
Arm/Group | Reactive Care (RC) | Proactive Care (PC)
Number analyzed (Participants) | 141 | 153
hours per night of CPAP use | 7.4 (2.2) | 6.3 (2.7)

2. Secondary Outcome: Change in Daytime Functioning at 6 and12 Weeks
Description: Change in daytime functioning will be measured using the Functional Outcomes of Sleep Quality (FOSQ) questionnaire. The FOSQ measures impact of sleepiness on activities of daily living (ADLs). The FOSQ-10 consists of 10 questions on a scale of 1 to 4 (1 = extreme difficulty, 4 = no difficulty). A lower score indicates more difficulty with ADLs due to lack of sleep. The FOSQ total score is the mean of subscale scores (ie, vigilance, productivity, social outcome, intimacy, activity) multiplied by 5. The scores range from 5 (maximum difficulty) to 20 (no difficulty). Change in FOSQ total score is calculated from baseline to end point, with higher (positive) values representing improvement. The worst possible change value would be -15 and the best would be +15.
Time Frame: 6 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reactive Care (RC) | Proactive Care (PC)
Number analyzed (Participants) | 141 | 153
score on a scale
  6 weeks | 15.2 (3.0) | 14.6 (3.7)
  12 weeks | 15.1 (3.2) | 14.6 (3.6)

3. Other Pre Specified Outcome: Change in Sleep Quality at 6 and 12 Weeks
Description: Change in sleep quality at 6 weeks and 12 weeks will be larger in the proactive care group compared to the reactive care group. This will be measured using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a self-rated, 19-item questionnaire used to assess sleep quality and disturbances over the previous 1 month. Items are scored on a Likert scale, with 0 being indicative of better sleep and the maximum value of 3 being indicative of poor sleep. PSQI scores can range from 0 to 21, with higher scores indicating worse sleep quality.
Time Frame: 6 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reactive Care (RC) | Proactive Care (PC)
Number analyzed (Participants) | 141 | 153
score on a scale
  6 weeks | 7.9 (4.1) | 8.8 (4.1)
  12 weeks | 7.6 (4.0) | 8.4 (4.1)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: An adverse event form was created for this project to assess/capture adverse events that may have been experienced as a result of being a participant in this study (e.g., adverse event type, adverse event date, adverse event description).
Arm/Group | Reactive Care (RC) | Proactive Care (PC)
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/153
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/153
Other Adverse Events (participants affected / at risk) | 0/141 | 0/153

LIMITATIONS AND CAVEATS:
The study utilized a national, electronic only recruitment method, which was primarily focused on the chronic obstructive pulmonary disease (COPD) and obstructive sleep apnea (OSA) communities. This may have resulted in a sample of participants who are more actively involved online seeking information and support for their medical condition.

Future studies would benefit from recruiting a more diverse sample of patients on a number of dimensions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT03446768/Prot_SAP_000.pdf